CLINICAL TRIAL: NCT01587885
Title: Protocol PT 11-29: Randomized, Open-label, Cross-over Pilot Study to Evaluate and Compare Two Omeprazole Containing Products for Relief of Frequent Heartburn
Brief Title: Comparison of Two Omeprazole-Containing Products for Relief of Frequent Heartburn (MK-0764A-036)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 18131; PT 11-29 (Other: Study Number); 0764A-036 (Other: Merck)
Record Dates: First submitted 2012-04-04; First posted 2012-04-30 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Heartburn
Keywords: Frequent Heartburn; Omeprazole; Omeprazole, sodium bicarbonate drug combination; Gastrointestinal Agents; Therapeutic Uses; Pharmacologic Actions; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action; Proton Pump Inhibitors
MeSH Terms: conditions — Heartburn | interventions — Omeprazole; Sodium Bicarbonate; omeprazole, sodium bicarbonate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omeprazole 20 mg + Sodium Bicarbonate 1100 mg (Experimental): Participants will receive omeprazole 20 mg + sodium bicarbonate 1100 mg once a day for 4 days, and then after a washout period, omeprazole 20 mg once a day for 4 days.
  Interventions: Drug: Omeprazole 20 mg + Sodium Bicarbonate 1100 mg; Drug: Omeprazole 20 mg
- Omeprazole 20 mg (Active Comparator): Participants will receive omeprazole 20 mg once a day for 4 days, and then after a washout period, omeprazole 20 mg + sodium bicarbonate 1100 mg once a day for 4 days.
  Interventions: Drug: Omeprazole 20 mg + Sodium Bicarbonate 1100 mg; Drug: Omeprazole 20 mg

INTERVENTIONS:
Drug: Omeprazole 20 mg + Sodium Bicarbonate 1100 mg — Capsules, orally
  Other Names: Zegerid™
Drug: Omeprazole 20 mg — Tablets, orally
  Other Names: Prilosec OTC™

SUMMARY:
This study will evaluate a single ingredient product (omeprazole 20 mg) with a combination product capsule (omeprazole 20 mg + sodium bicarbonate 1100 mg) in participants with frequent heartburn.

ELIGIBILITY:
Inclusion Criteria:

* Females of reproductive potential must demonstrate a negative urine pregnancy test and agree to use an acceptable method of birth control
* Suffer from frequent heartburn
* Refrain from taking non-study medicine or treatment for heartburn for the duration of the study
* Be free of any clinically significant disease that requires a physician's care
* Read and understand English

Exclusion Criteria:

* Any significant medical condition which is a contraindication to the use of omeprazole or sodium bicarbonate
* Known hypersensitivity to the study drugs or any components
* Experiencing any of the following: trouble or pain with swallowing food, vomiting with blood, bloody or black stools
* Participation in another investigational study within 4 weeks prior to the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Omeprazole 20mg+Sodium Bicarbonate 1100mg Then Omeprazole 20mg: Participants will receive omeprazole 20 mg + sodium bicarbonate 1100 mg once a day for 4 days, and then after a washout period, omeprazole 20 mg once a day for 4 days.
- Omeprazole 20mg Then Omeprazole 20mg+Sodium Bicarbonate 1100mg: Participants will receive omeprazole 20 mg once a day for 4 days, and then after a washout period, omeprazole 20 mg + sodium bicarbonate 1100 mg once a day for 4 days.
Period: Treatment Period 1
Arm/Group | Omeprazole 20mg+Sodium Bicarbonate 1100mg Then Omeprazole 20mg | Omeprazole 20mg Then Omeprazole 20mg+Sodium Bicarbonate 1100mg
Started | 26 | 22
Completed | 26 | 19
Not Completed | 0 | 3
Not completed — Failure to Return | 0 | 1
Not completed — Protocol Violation | 0 | 2
Period: Treatment Period 2
Arm/Group | Omeprazole 20mg+Sodium Bicarbonate 1100mg Then Omeprazole 20mg | Omeprazole 20mg Then Omeprazole 20mg+Sodium Bicarbonate 1100mg
Started | 26 | 19
Completed | 26 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who were randomized and received study drug.
Arm/Group | All Participants
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (12.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Time-to-onset of Heartburn Relief
Description: Time-to-onset of heartburn relief was defined as earliest time following start of treatment that participant experienced a reduction of at least one grade from baseline in the severity of heartburn. Severity of heartburn was evaluated by the participant using the 4-point Likert Scale, which rated heartburn severity as follows:
  Absent (0): Heartburn is not present.
  Mild (1): Heartburn did not last long or was easily tolerated.
  Moderate (2): Heartburn caused discomfort and interrupted usual activities.
  Severe (3): Heartburn caused great interference with usual activities and may have been incapacitating.
Time Frame: Start of treatment until onset of heartburn relief, up to 24 hours
Population: Participants in the modified Intent-to-Treat (mITT) population, consisting of all randomized participants who received study drug and who provided efficacy data for at least one of the study drugs for the variable and time point analyzed.
  One participant completed the study but the participant's data was corrupted and therefore not included.
Measure: Median (Inter-Quartile Range); unit: Minutes
Groups:
- Omeprazole 20 mg + Sodium Bicarbonate 1100 mg: Participants will receive omeprazole 20 mg + sodium bicarbonate 1100 mg once a day for 4 days.
- Omeprazole 20 mg: Participants will receive omeprazole 20 mg once a day for 4 days.
Arm/Group | Omeprazole 20 mg + Sodium Bicarbonate 1100 mg | Omeprazole 20 mg
Number analyzed (Participants) | 44 | 44
Minutes | 30.0 [30.0 to 75.0] | 60.0 [30.0 to 105.0]
Statistical Analysis 1: Comparison: Omeprazole 20 mg + Sodium Bicarbonate 1100 mg vs Omeprazole 20 mg; Test type: Superiority or Other; p < 0.0480, Regression, Cox; Hazard Ratio (HR) = 1.548

2. Secondary Outcome: Percentage of Participants Experiencing Onset and Demonstrating Duration of Heartburn Relief Over Time
Description: Onset of heartburn relief was defined as a reduction of at least one grade from baseline in the severity of heartburn following start of treatment. Severity of heartburn was evaluated by the participant using the 4-point Likert Scale, which rated heartburn severity as follows:
  Absent (0): Heartburn is not present.
  Mild (1): Heartburn did not last long or was easily tolerated.
  Moderate (2): Heartburn caused discomfort and interrupted usual activities.
  Severe (3): Heartburn caused great interference with usual activities and may have been incapacitating.
Time Frame: Start of treatment until onset of heartburn relief, up to 72 hours
Population: Participants in the mITT population, consisting of all randomized participants who received study drug and who provided efficacy data for at least one of the study drugs for the variable and time point analyzed.
  One participant completed the study but the participant's data was corrupted and therefore not included.
Measure: Number; unit: percentage of participants
Arm/Group | Omeprazole 20 mg + Sodium Bicarbonate 1100 mg | Omeprazole 20 mg
Number analyzed (Participants) | 44 | 44
percentage of participants
  ≤15 minutes | 20.5 | 13.6
  ≤30 minutes | 52.3 | 27.3
  ≤60 minutes | 75.0 | 61.4
  ≤90 minutes | 90.9 | 75.0
  ≤120 minutes | 95.5 | 88.6
  ≤180 minutes | 100.0 | 90.9
  ≤1440 minutes (24 hours) | 100.0 | 93.2
  ≤2880 minutes (48 hours) | 100.0 | 95.5
  ≤4320 minutes (72 hours) | 100.0 | 100.0

3. Secondary Outcome: Number of Participants Preferring Each Treatment for Heartburn Control: Final Subjective Questionnaire
Description: Participants completed a Final Subjective Questionnaire for Treatment Preference. Question 1 asked participants to compare the 2 treatments for Heartburn Control.
Time Frame: At end of study (approx. Study Day 40)
Population: Participants in the Intent-to-Treat (ITT) population, consisting of all participants who were randomized, took study medication at the beginning of treatment period 1, and provided data.
Measure: Number; unit: participants
Arm/Group | All Treated Participants
Number analyzed (Participants) | 48
participants
  Preferred omeprazole+sodium bicarbonate | 14
  Preferred omeprazole | 17
  Preferred both equally | 9
  Missing data | 8

4. Secondary Outcome: Number of Participants Preferring Each Treatment for Heartburn Relief: Final Subjective Questionnaire
Description: Participants completed a Final Subjective Questionnaire for Treatment Preference. Question 2 asked participants to compare the 2 treatments for Heartburn Relief.
Time Frame: At end of study (approx. Study Day 40)
Population: Participants in the ITT population, consisting of all participants who were randomized, took study medication at the beginning of treatment period 1, and provided data.
Measure: Number; unit: participants
Arm/Group | All Treated Participants
Number analyzed (Participants) | 48
participants
  Preferred omeprazole+sodium bicarbonate | 16
  Preferred omeprazole | 16
  Preferred both equally | 7
  Preferred neither | 1
  Missing data | 8

5. Secondary Outcome: Number of Participants Preferring Each Treatment Overall: Final Subjective Questionnaire
Description: Participants completed a Final Subjective Questionnaire for Treatment Preference. Question 3 asked participants to compare the 2 treatments for their overall preference.
Time Frame: At end of study (approx. Study Day 40)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | All Treated Participants
Number analyzed (Participants) | 48
participants
  Preferred omeprazole+sodium bicarbonate | 17
  Preferred omeprazole | 17
  Preferred both equally | 6
  Missing data | 8

6. Secondary Outcome: Percentage of Participants Affected By Heartburn Symptoms: End of Treatment Quality of Life Questionnaire
Description: End of Treatment Quality of Life was based on a questionnaire regarding quality-of-life issues associated with heartburn, completed by participants at the end of treatment period 1 and the end of treatment period 2.
Time Frame: End of treatment period 1 and end of treatment period 2
Population: Participants in the mITT population, consisting of all randomized participants who received study drug and who provided efficacy data for at least one of the study drugs for the variable and time point analyzed.
Measure: Number; unit: percentage of partcipants
Arm/Group | Omeprazole 20 mg + Sodium Bicarbonate 1100 mg | Omeprazole 20 mg
Number analyzed (Participants) | 40 | 40
percentage of partcipants
  heartburn symptoms affected daily activities | 30.0 | 30.0
  heartburn symtoms caused trouble falling asleep | 27.5 | 25.0
  heartburn symptoms awoke participant | 22.5 | 32.5
  slept on incline due to heartburn symptoms | 35.0 | 47.5
  medicine helped with full night's rest | 90.0 | 95.0

ADVERSE EVENTS:
Description: Three participants discontinued the study prior to receiving Omeprazole 20 mg + Sodium Bicarbonate 1100 mg. Therefore, only 45 participants received Omeprazole 20 mg + Sodium Bicarbonate 1100 mg.
Arm/Group | Omeprazole 20 mg + Sodium Bicarbonate 1100 mg | Omeprazole 20 mg
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/48
Other Adverse Events (participants affected / at risk) | 0/45 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MERCK retains the title to and exclusive right to publish all documentation, research data, records, raw data, other work product, data, and/or results generated with respect to the Services and/or the Study ("Work Product"). Such Work Product will be retained in the CRO archive in compliance with regulatory requirements.